CLINICAL TRIAL: NCT05078164
Title: Preventing Firearm Violence in Youth: A Hospital-based Prevention Strategy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20022975; 1R01HD108025 (NIH)
Record Dates: First submitted 2021-09-29; First posted 2021-10-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Violence in Adolescence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Youth who will not receive BTG services and will receive treatment as usual (TAU) in the hospital.
- Bridging the Gap (BTG) (Experimental): Youth randomized to Bridging the Gap (BTG) services will receive a hospital-based violence prevention program with 3-months of community case management and a firearm counseling program.
  Interventions: Behavioral: Bridging the Gap (BTG)

INTERVENTIONS:
Behavioral: Bridging the Gap (BTG) — Bridging the Gap: Bridging the Gap is a hybrid model for violence prevention which integrates a hospital-based brief violence intervention (BVI) delivered to the patient while in hospital with a wrap-around community case management prevention strategy.
  Firearm Counseling Program: The firearm counseling program was developed to be administered in the hospital alongside the 6-step intervention program, as well as in the patient's home after hospital discharge. The firearm safety counseling program includes 3 components aimed at understanding patient risk, reducing firearm-related violence risk-factors, and helping patients increase firearm safety practices.
  Arms: Bridging the Gap (BTG)

SUMMARY:
The goal of the study is to understand if hospital-based violence interventions are effective for reducing youth violence among violently injured youth. This study will allow researchers to learn more about the intervention's effectiveness. The researchers also want to understand if the violence intervention impacts other behaviors, such as firearm use, drug use, aggression, risky behaviors, and rates of violent re-injury.

DETAILED DESCRIPTION:
The purpose of this research study is to find out if a hospital-based violence intervention (Bridging the Gap) is effective for reducing youth violence. Researchers think that youth who receive the Bridging the Gap will see greater improvements than youth who do not receive the intervention. Approximately 300 youth patients and 300 adult caregivers will enroll in this study. Participants will be randomized into a study group (either Bridging the Gap or Treatment as Usual). If patients agree to the study but do not like the group they are assigned to, they can request to switch groups. Participants assigned to the Treatment as Usual intervention will receive a brief violence awareness brochure during their hospital stay. Participants assigned to the Bridging the Gap intervention will receive an in-hospital intervention and, once released from the hospital, will receive 3-months of community case management services with their families. The study team thinks that youth who receive the Bridging the Gap intervention will see greater improvements than youth who do not receive the intervention. Participation in this study will last up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Youth are aged 10-17 years and their adult caregivers are aged 18 years and older
2. Receiving treatment in the hospital for a violence-related injury (e.g., gunshot wound) or referred to BTG/IVPP services
3. English speaking
4. Eligible for BTG services (which includes living within the BTG catchment area for the hospital; Richmond City and neighboring counties)

Exclusion Criteria:

1. Youth are < 10 years old
2. Youth are > 18 years old
3. Prisoners

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Firearm-related violence | 6 months
  Total number of unique firearm-related violence incidents will be assessed multiple ways including self-report assessment and semi-structured clinical assessments.
Firearm-related carrying behaviors | 6 months
  Total number of firearm-related carrying behaviors will be assessed multiple ways including self-report assessment and semi-structured clinical assessments.
Firearm-related beliefs | 6 months
  Total number of firearm-related beliefs endorsed will be assessed multiple ways including self-report assessment and semi-structured clinical assessments.
Firearm-related re-injury | 6 months
  Total number of unique firearm-related re-injury incidents will be measured multiple ways including self-report, caregiver-report, hospital records, and the National Death Index.
Firearm-related mortality | 6 months
  Number of deaths will be collected from hospital records and the National Death Index.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Thomson, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No